CLINICAL TRIAL: NCT04730765
Title: Assesment of Quality of Life and Digestive and Genitourinary Functional Sequelae After Elective Left Colectomy for Sigmoid Diverticulitis. National Multicenter Prospective Observational Study
Brief Title: Quality of Life (QOL) After Elective Sigmoidectomy for Diverticular Diseases (DIVERTI)
Acronym: DIVERTI-QDV
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Caen (Other)
Collaborators: Association Francaise de Chirurgie (Other)
Responsible Party: Sponsor
Other Study IDs: 20-181; 2020-A02802-37 (Other: IDRCB Number)
Record Dates: First submitted 2021-01-26; First posted 2021-01-29 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-03

CONDITIONS: Diverticular Disease of Left Side of Colon
Keywords: Quality Of Life; Elective colectomy; Diverticular diseases
MeSH Terms: conditions — Diverticular Diseases | interventions — Anti-Infective Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgical Experimental Group: Patient operated between 01/02/2021 and 30/07/2021, in elective situation of sigmoid diverticulitis
  Interventions: Procedure: left elective colectomy (Surgical Experimental Group)
- Medical Control Group: Patient not operated and medically treated
  Interventions: Drug: antibiotic therapy (medical Control Group)

INTERVENTIONS:
Procedure: left elective colectomy (Surgical Experimental Group) — Conventional laparoscopic resection of the sigmoid colon is performed using four ports. The left colon is mobilised from the lateral side along Gerota's fascia. The splenic flexure is mobilised at the discretion of surgeons. The mesentery of the sigmoid colon is then medially fenestrated at the promontory level. The superior rectal artery as well as the inferior mesenteric artery and vein are identified and are cut using tissue-sealing devices. A linear stapler device is applied for division of the large intestine. The sigmoid is retracted through a Pfannenstiel incision or enlargement of the left lower abdominal incision. Colorectal anastomosis is performed using a double stapling technique following open resection of the affected colon.
  Groups: Surgical Experimental Group
Drug: antibiotic therapy (medical Control Group) — Antibiotic treatement for 10 days by oral or intravenous administration
  Groups: Medical Control Group

SUMMARY:
Acute diverticulitis of the left colon is among the most common abdominal disorders. To date, both conservative therapy in uncomplicated stages and emergency surgery in perforated disease with peritonitis are consensual. The best treatment strategy for other situations (i.e., smoldering, healed abscesses, recurrences) is still under debate. On the other hand, the best treatment strategy for complicated disease as well as for recurrent stages is still under debate. In these cases, elective surgery can be proposed on a case-by-case basis. Current French guideline recommendations have been updated in 2017. In theory, the objective of elective surgical treatment is to prevent the recurrence and/or complication of the diverticulitis, that might lead to the creation of a stoma. In France, nearly 12,000 prophylactic colectomies for diverticulitis are performed per year. Importantly, elective surgical treatment is associated with the relevant intrinsic morbidity (9.6% major complications within the Sigma Trial), the potential need for unplanned stoma formation of 1%-14% and a significant risk of persisting postoperative complaints. Up to 25% of patients who have undergone a scheduled sigmoid colectomy suffer from ongoing abdominal symptoms. Levack et al found the risk of faecal incontinence to be 24.8% after a sigmoidectomy. Moreover, faecal urgency occurred in 19.6% of patients, and incompleteness of emptying occurred in 20.8%., altering their quality of life (QOL).

To out knowledge, few data are available in the literature concerning the evaluation of QOL after elective sigmoid colectomy. Although QOL was significantly improved after surgery compared to conservative medical treatment, these results were questionable due to the heterogeneity of the studies and the lack of direct comparison of the two therapeutic approaches. Only one recent randomized study reported similar results but this one was prematurely stopped due to inclusion difficulties. The evaluation of digestive and genitourinary functional sequelae is based only on short series, most often retrospective. In summary, evidence on disease-specific characteristics influencing postoperative quality of life is lacking.

The aim of this prospective multicenter study is : (i) to evaluate the QOL and functional sequelae at 6 and 12 months in patients operated on for elective left colectomy and, (ii) to compare them to a population of non-operating diverticulitis patients.

DETAILED DESCRIPTION:
Design The DIVERTI-QOL study is a prospective, multicentre, and observational study. The study will start in February 2021. Recruitment will be completed in July 2021. Overall, the inclusion of 110 patients in each arm is planned. 37 french hospitals agreed to participate in this study.

Allocation for surgery

The allocation to conservative or surgical therapy will be performed at the inclusion in the study. Possible indications for surgery are listed below :

* Persisting abdominal complaints (smouldering diverticular disease) after uncomplicated diverticulitis (Classification of Diverticular Disease (CDD) Stage 1, modified Hinchey 0+Ia).
* Persisting abdominal complaints after covered perforation and/or pericolic 'microabscesses' (1cm) (CDD Stage 2b).
* Chronic or recurrent diverticulitis with persisting abdominal complaints
* diverticulitis complicated by an abscess >1 cm
* divericulitisin a patient requiring long-term immunosuppressive therapy (with the exception of a neoplastic disease undergoing treatment)

ELIGIBILITY:
inclusion criteria:

* Patient who has received informed information and has not expressed opposition to participation
* Francophone patient
* Patient affiliated to a social security or equivalent system
* Patient taken in charge for :

  * smoldering DS after DS Hinchey I
  * persistence of symptoms after DS complicated by a peri-sigmoid abscess <1cm with resolution of inflammation
  * DS complicated with an abscess >1cm (Hinchey II)
  * Recurrent episodes of DS
  * DS in a patient requiring long-term immunosuppressive therapy (except for neoplastic disease undergoing treatment)
* Patient operated between 01/02/2021 and 30/07/2021, in elective situation of sigmoid diverticulitis (surgical experimental group) or patient not operated and medically treated (medical control group)

Exclusion Criteria:

Subjects meeting only one of the following non-inclusion criteria may not be eligible to participate in the research:

* Patient who is a minor or over 70 years of age
* Patient undergoing emergency surgery for sigmoid diverticulitis due to a complication (peritonitis, hemorrhage, failure of drainage diverticular abscess)
* diverticulitis complicated by fistula and/or symptomatic stenosis
* Colorectal resection protected by an ostomy or Hartmann's intervention
* Discovery of colorectal cancer on the operating room
* Patient operated on for diverticulitis of the right colon
* Neoplastic disease under treatment and/or evolving

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The allocation to conservative or surgical therapy will be performed at the inclusion in the study. Possible indications for surgery are listed below :
  * Persisting abdominal complaints (smouldering diverticular disease) after uncomplicated diverticulitis (Classification of Diverticular Disease (CDD) Stage 1, modified Hinchey 0+Ia).
  * Persisting abdominal complaints after covered perforation and/or pericolic 'microabscesses' (1cm) (CDD Stage 2b).
  * Chronic or recurrent diverticulitis with persisting abdominal complaints
  * diverticulitis complicated by an abscess >1 cm
  * divericulitisin a patient requiring long-term immunosuppressive therapy (with the exception of a neoplastic disease undergoing treatment)
Sampling Method: Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2021-09-15 (Estimated); Primary Completion 2021-10-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative HrQoL 6months postoperatively; quality of life will be measured by the Gastrointestinal Quality of Life Index (GIQLI) | 6 months
  The score consists of 36 questions or items rated from 0 to 4 (0 being the worst and 4 the best). The sum of the scores constitutes the overall quality of life score; the ideal score is 144. The items cover 5 dimensions or sub-scales: symptoms (19 items), physical condition (7 items), emotions (5 items), social integration (4 items) and the effect of medical or surgical treatment (1 item). The questionnaire is considered usable if the missing data do not concern more than 2 questions. The QOL score (global and sub-scales) is calculated for all complete answers.
  36 questions

SECONDARY OUTCOMES:
Health-related QOL will also be assessed according to the 5 dimensions of the GIQLI but also using the EQ-5D-5L score. The EuroQdV 5-Dimensions 5-Level (EQ-5D-5L) | 6 and 12 months
  The EuroQdV 5-Dimensional 5-Level (EQ-5D-5L) is a widely used utility instrument. Its descriptive system consists of five questions that cover the dimensions of mobility, personal autonomy, daily activities, pain/comfort, anxiety/depression, each with five possible answers that qualitatively reflect the presence of a problem (no problem, mild, moderate, severe and extreme).
Hostoperative HrQoL 12months postoperatively; quality of life will be measured by the Gastrointestinal Quality of Life Index (GIQLI) | 12 months
  The score consists of 36 questions or items rated from 0 to 4 (0 being the worst and 4 the best). The sum of the scores constitutes the overall quality of life score; the ideal score is 144. The items cover 5 dimensions or sub-scales: symptoms (19 items), physical condition (7 items), emotions (5 items), social integration (4 items) and the effect of medical or surgical treatment (1 item). The questionnaire is considered usable if the missing data do not concern more than 2 questions. The QOL score (global and sub-scales) is calculated for all complete answers.
  36 questions
Digestive sequelae will be assessed using the LARS score, the French version of which is currently being validated, genitourinary sequelae will be assessed using a simplified questionnaire. | 6 and 12 months
  The LARS score developed and validated in Denmark includes 5 items: gas incontinence, liquid stool incontinence, fragmentation and urgency (specifying for each item the frequency: never, less than once a week or more than once a week) and stool frequency (specifying respectively more than 7, between 4 and 7, between 1 and 3 and less than one stool per 24 hours). It assesses how these functional digestive sequelae affect QOL, i.e. never, very little, often or all the time. There is no Prior Resection Syndrome (PRS) if the score is between 0 and 20, but there is a minor PRS if the score is between 21 and 29 and a major PRS if the score is between 30 and 42.
Morbidity and mortality at 90 days will be assessed using the International Classification of Dindo-Clavian Disease and by follow-up | 90 days
  Grade I Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions Allowed therapeutic regimens are: drugs as antiemetics, antipyretics, analgetics, diuretics and electrolytes and physiotherapy. This grade also includes wound infections opened at the bedside.
  Grade II Requiring pharmacological treatment with drugs other than such allowed for grade I complications.
  Blood transfusionsand total parenteral nutritionare also included. Grade III Requiring surgical, endoscopic or radiological intervention
  * IIIa Intervention not under general anesthesia
  * IIIb Intervention under general anesthesia Grade IV Life-threatening complication (including CNS complications)* requiring IC/ICU-management
  * IVa single organ dysfunction (including dialysis)
  * IVb multiorgandysfunction Grade V Death of a patient

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bolkenstein HE, Consten ECJ, van der Palen J, van de Wall BJM, Broeders IAMJ, Bemelman WA, Lange JF, Boermeester MA, Draaisma WA; Dutch Diverticular Disease (3D) Collaborative Study Group. Long-term Outcome of Surgery Versus Conservative Management for Recurrent and Ongoing Complaints After an Episode of Diverticulitis: 5-year Follow-up Results of a Multicenter Randomized Controlled Trial (DIRECT-Trial). Ann Surg. 2019 Apr;269(4):612-620. doi: 10.1097/SLA.0000000000003033. PMID 30247329
- [Result] Forgione A, Guraya SY. Elective colonic resection after acute diverticulitis improves quality of life, intestinal symptoms and functional outcome: experts' perspectives and review of literature. Updates Surg. 2016 Mar;68(1):53-8. doi: 10.1007/s13304-016-0349-0. Epub 2016 Mar 25. PMID 27015932
- [Result] Schultz JK, Azhar N, Binda GA, Barbara G, Biondo S, Boermeester MA, Chabok A, Consten ECJ, van Dijk ST, Johanssen A, Kruis W, Lambrichts D, Post S, Ris F, Rockall TA, Samuelsson A, Di Saverio S, Tartaglia D, Thorisson A, Winter DC, Bemelman W, Angenete E. European Society of Coloproctology: guidelines for the management of diverticular disease of the colon. Colorectal Dis. 2020 Sep;22 Suppl 2:5-28. doi: 10.1111/codi.15140. Epub 2020 Jul 7. PMID 32638537
- [Result] Sohn M, Agha A, Iesalnieks I, Bremer S, Trum S, Di Cerbo F, Nerlich A, Lotz N, Klieser E, Hochrein A, Schredl P, Kalcheva D, Emmanuel K, Presl J. PREDICtors for health-related quality of life after elective sigmoidectomy for DIVerticular disease: the PREDIC-DIV study protocol of a prospective multicentric transnational observational study. BMJ Open. 2020 Mar 24;10(3):e034385. doi: 10.1136/bmjopen-2019-034385. PMID 32209628